CLINICAL TRIAL: NCT02772003
Title: Phase I Trial of a Therapeutic DNA Vaccine for Chronic Hepatitis C Virus (HCV) Infection
Brief Title: DNA Vaccine Therapy in Treating Patients With Chronic Hepatitis C Virus Infection
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Inovio Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: NCI-2015-00558; NCI-2015-00558 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HHSN261201200042I; N01-CN-2012-00042; MAY2013-02-01 (Other: Mayo Clinic in Rochester); MAY2013-02-01 (Other: DCP); N01CN00042 (NIH); P30CA015083 (NIH); NCT02822079 (obsolete NCT alias)
Record Dates: First submitted 2016-04-27; First posted 2016-05-13 (Estimated); Last update posted 2026-02-12 (Actual); Status verified 2025-09

CONDITIONS: Chronic Hepatitis; Hepatitis C Infection; Hepatocellular Carcinoma
MeSH Terms: conditions — Hepatitis, Chronic; Hepatitis C; Carcinoma, Hepatocellular | interventions — rocakinogene sifuplasmid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (INO-8000, INO-9012, EP) (Experimental): Patients receive INO-8000 IM and DNA plasmid encoding interleukin-12 INO-9012 IM (dose levels 2-4) followed by EP at day 0 and at weeks 4, 12, and 24.
  Interventions: Biological: Electroporation-Mediated Plasmid DNA Vaccine Therapy; Biological: HCV DNA Vaccine INO-8000; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Biological: Rocakinogene Sifuplasmid

INTERVENTIONS:
Biological: Electroporation-Mediated Plasmid DNA Vaccine Therapy — Undergo electroporation
Biological: HCV DNA Vaccine INO-8000 — Given IM
  Other Names: INO-8000
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Biological: Rocakinogene Sifuplasmid — Given IM
  Other Names: DNA Plasmid Encoding Interleukin-12 INO-9012; INO-9012

SUMMARY:
This phase I trial studies the side effects and best dose of deoxyribonucleic acid (DNA) vaccine therapy in treating patients with hepatitis C virus (HCV) infection that persists or progresses over a long period of time. Vaccines made from DNA may help the body build an effective immune response to kill cancer cells that express HCV infection.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety profile of the HCV DNA vaccine, consisting of INO-8000 (HCV antigen DNA) alone or co-administered with INO-9012 (interleukin [IL]-12 adjuvant DNA) (DNA plasmid encoding interleukin-12 INO-9012).

II. To identify a dose of INO-9012 (IL-12 adjuvant DNA) for co-administration with INO-8000 (HCV antigen DNA) based on induction of HCV-specific interferon (IFN)-gamma production by peripheral blood mononuclear cells at 26 weeks compared to baseline in HCV-infected participants.

TRANSLATIONAL OBJECTIVES:

I. Determine the rate at which INO-8000 with different doses of INO-9012 induces a > 1 log decrease (or undetectable) in HCV ribonucleic acid (RNA) level at weeks 14 and 26.

II. Determine the rate at which INO-8000 with different doses of INO-9012 induces an end-of-treatment undetectable HCV RNA (end-of-treatment virologic response - EVR) at 26 weeks and a sustained virologic response (SVR) at 36 weeks.

III. Determine the rate at which INO-8000 with different doses of INO-9012 induces other parameters of cluster of differentiation (CD)8 and CD4 T lymphocyte responses as measured by flow cytometry, and antibody responses to HCV antigen at weeks 14 and 26.

OUTLINE: This is a dose-escalation study of INO-9012.

Patients receive INO-8000 intramuscularly (IM) and DNA plasmid encoding interleukin-12 INO-9012 IM (dose levels 2-4) followed by electroporation (EP) at day 0 and at weeks 4, 12, and 24.

After completion of study treatment, patients are followed up at weeks 48 and 76.

ELIGIBILITY:
Inclusion Criteria:

* PRE-REGISTRATION INCLUSION CRITERIA
* Presence of active, chronic HCV infection confirmed by positive HCV RNA
* Willingness to use adequate contraception to avoid pregnancy or impregnation for the duration of study participation; Note:

  * The effects of INO-8000 with or without INO-9012 on the developing human fetus at the recommended therapeutic dose are unknown; for this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation
  * For men and women who are not postmenopausal (i.e., >= 12 months of non-therapy-induced amenorrhea, confirmed by follicle stimulating hormone [FSH], if not on hormone replacement) or surgically sterile (vasectomy in males or absence of ovaries and/or uterus in females), agreement to remain abstinent or use highly effective or combined contraceptive methods that result in a failure rate of < 1% per year during the treatment period and at least through week 12 after last dose
  * Abstinence is only acceptable if it is in line with the preferred and usual lifestyle of the subject; periodic abstinence (e.g., calendar, ovulation, symptothermal, or post-ovulation methods) and withdrawal are not acceptable methods of contraception
  * Examples of contraceptive methods with an expected failure rate of < 1% per year include male sterilization and hormonal implants; alternatively, proper use of combined oral or injected hormonal contraceptives and certain intrauterine devices or two methods (e.g., two barrier methods such as a condom and a cervical cap) may be combined to achieve a failure rate of < 1% per year (barrier methods must always be supplemented with the use of a spermicide)
  * Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately
  * Should a female partner of a male study participant become pregnant while the male participant is on study, the male participant should inform his study physician immediately
* Willingness to avoid excessive use of alcohol during the study; note: excessive use is defined as drinking >= 8 alcoholic drinks per week on average
* Willingness to provide blood samples for research tests specified in the protocol
* Ability to understand and willingness to sign a written informed consent document
* REGISTRATION INCLUSION CRITERIA
* Serum or plasma HCV RNA level >= 10,000 IU/mL
* Screening HCV genotype, demonstrating genotype 1
* Alpha feto protein (AFP) levels within normal institutional limits or judged to be not clinically significant by the investigator; Exception: If deemed clinically significant, then liver imaging must be available within previous 6 months (e.g., ultrasound, computed tomography [CT] scan, magnetic resonance imaging [MRI]) showing no evidence of hepatocellular carcinoma
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Screening laboratory values (serum chemistry, hematology, prothrombin time [PT](international normalized ratio [INR])/activated partial thromboplastin time [APTT], and creatine phosphokinase [CPK]) obtained up to 45 days prior to administration of first vaccine injection on day 0 within institutional normal range or judged to be not clinically significant by principal investigator (PI) and medical monitor
* 12-lead electrocardiogram (ECG) showing normal heart rhythm; note: if there are abnormalities, then the abnormalities must be deemed of no clinical significance

Exclusion Criteria:

* PRE-REGISTRATION EXCLUSION CRITERIA
* Failure of previous HCV therapies
* Human immunodeficiency virus (HIV) infection
* Any previous treatment for HCV =< 6 months prior to registration
* Other uncontrolled immune-compromising illness
* Autoimmune disorders, transplant recipients, other immunosuppression including any concurrent condition requiring the use of immunosuppressive/ immunomodulating agents; Exception: eye drop-containing and infrequent inhaled corticosteroids are permissible; topical corticosteroids are permissible at locations other than the administration site (upper arm); Note: All systemic corticosteroids must be discontinued at least 4 weeks prior to randomization; inhaled corticosteroids must be discontinued >= 48 hours prior to randomization and courses of more than 2 weeks are not permissible within 4 weeks of randomization
* Ongoing hepatitis B virus (HBV) infection
* Documented evidence of fibrosis or cirrhosis (Metavir 2, 3, and 4) and subjects with significant extrahepatic manifestations of hepatitis C (such as cryoglobulinemia with symptoms or evidence of end-organ manifestations, renal disease, type 2 diabetes, or porphyria cutanea tarda
* Other known causes of significant liver disease including chronic or acute hepatitis B, acute hepatitis A, hemochromatosis, or homozygote alpha-1 antitrypsin deficiency
* Active malignancy; exception: non-melanoma skin cancers cancer(s) for which diagnosis and treatment was completed >= 3 years prior to pre-registration
* History of major organ transplantation with an existing functional graft
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* History of cardiac arrhythmia, controlled or uncontrolled, including ventricular and supraventricular arrhythmia
* Pregnant or nursing women; Note: Pregnant women are excluded from this study because INO-8000 has an unknown potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with this DNA vaccine, breastfeeding should be discontinued if the mother is treated with INO-8000
* Current diagnosis or history of cardiac pre-excitation syndromes (e.g. Wolff-Parkinson-White)
* Metal implants on same limb as intended administration site
* Tattoos, scars, active lesions, or rashes =< 2 cm of the intended site of study treatment
* Documentation of history of seizure within previous 5 years
* Pacemaker or other implanted device
* Any condition that, in the clinical judgement of the investigator, would place a participant at unreasonably increased risk
* REGISTRATION EXCLUSION CRITERIA
* Receiving any other investigational agents =< 6 months prior to Registration
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to INO-8000 and INO-9012

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-06-06 (Actual); Primary Completion 2020-03-04 (Actual); Study Completion 2026-03-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity | Baseline to 26 weeks
  Will be defined as an adverse event occurring after the initial vaccine administration, based on the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0. The percentage of participants who experience grade 3 or worse adverse events and administration-site reactions following each dose will be summarized using descriptive statistics across each dose level.
Mean change of interferon-gamma production by peripheral blood mononuclear cells | Baseline to 26 weeks
  Change in production of interferon-gamma by peripheral blood mononuclear cells will be based on a one-way analysis of variance model using data from all dose levels at the 2-sided 5% level. Mean change (and % change) and the associated 95% confidence intervals in the production of IFN-gamma by peripheral blood mononuclear cells for all evaluable participants enrolled at each dose level will be computed, and compared across the dose levels in an exploratory fashion using graphical approaches, one-way analysis of variance models etc. to ascertain a dose-response curve.

OTHER OUTCOMES:
Percentage of participants with > 1 log decrease (or undetectable) in hepatitis C virus ribonucleic acid level | Up to 26 weeks
  The point estimate (and the associated 95% confidence intervals) for primary immune response endpoint will be estimated within each arm and formally compared using a chi-squared test (or Fisher's exact test, if the data warrant). A logistic regression analysis will also be utilized to adjust for potential baseline covariates considered critical for this population.
Percentage of participants with end-of-treatment undetectable hepatitis C virus ribonucleic acid for the dose levels determined to be safe | 26 weeks
  The immune response comparisons will be made using descriptive statistics and graphical methods for both phases of the study. Descriptive statistics and simple scatter plots will be generated to review the continuous immune response data. For continuous immune response values, the actual and % change in the level of each of the biomarkers from baseline to post-baseline time points will be explored within each dose level/arm using Wilcoxon signed rank tests, and paired sample t-tests.
Sustained virologic response defined as undetectable hepatitis C virus ribonucleic acid | 36 weeks
  The immune response comparisons will be made using descriptive statistics and graphical methods for both phases of the study. Descriptive statistics and simple scatter plots will be generated to review the continuous immune response data. For continuous immune response values, the actual and % change in the level of each of the biomarkers from baseline to post-baseline time points will be explored within each dose level/arm using Wilcoxon signed rank tests, and paired sample t-tests.
CD8 and CD4 T lymphocyte responses as measured by flow cytometry, and antibody responses, to hepatitis C virus antigen for the dose levels determined to be safe | Up to 26 weeks
  The immune response comparisons will be made using descriptive statistics and graphical methods for both phases of the study. Descriptive statistics and simple scatter plots will be generated to review the continuous immune response data. For continuous immune response values, the actual and % change in the level of each of the biomarkers from baseline to post-baseline time points will be explored within each dose level/arm using Wilcoxon signed rank tests, and paired sample t-tests.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey M Jacobson, Principal Investigator — Mayo Clinic
Locations (5):
- United States (4):
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Case Western Reserve University, Cleveland, Ohio
  - Temple University Hospital, Philadelphia, Pennsylvania
- University of Puerto Rico, San Juan, Puerto Rico